CLINICAL TRIAL: NCT02184052
Title: Meloxicam (MOBIC®) Ampoule Post Marketing Surveillance Study
Brief Title: Safety and Efficacy of Mobic® Ampoules in the Initiation of Treatment of Painful Exacerbations of Osteoarthritis, Rheumatoid Arthritis and Other Similar Painful Inflammatory Conditions
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 107.267
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meloxicam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Meloxicam
  Interventions: Drug: Meloxicam

INTERVENTIONS:
Drug: Meloxicam — 7.5 mg or 15 mg

SUMMARY:
Study to determine the safety and efficacy of Mobic® ampoules in the initiation of treatment of painful exacerbations of osteoarthritis, rheumatoid arthritis and other similar painful inflammatory conditions.

ELIGIBILITY:
Inclusion Criteria:

* Painful acute exacerbations of inflammatory rheumatism (rheumatoid arthritis and ankylosing spondylitis), painful acute exacerbations of osteoarthritis and other similar conditions requiring acute treatment with an anti-inflammatory drug

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2003-07; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Overall assessment of degree of pain on a 3-point scale | up to 3 days

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 3 days